CLINICAL TRIAL: NCT04419350
Title: Microneedling for Acquired Hypomelanosis : A Randomized Controlled Trial
Brief Title: Microneedling for Acquired Hypomelanosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Julbahar Ibrahim, Dermatology resident,Principal investigator-Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MN for acquired hypomelanosis
Record Dates: First submitted 2020-05-23; First posted 2020-06-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Acquired Hypomelanosis
Keywords: Microneedling; Dermaroller; acquired hypomelanosis; skin pigmentation; hypopigmentation; patient satisfaction; leukoderma
MeSH Terms: conditions — Pigmentation Disorders; Hypopigmentation; Patient Satisfaction; Vitiligo | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: * The area to be treated will be specified and split into two halves then randomized using sealed envelope into one of both arms: treatment or no treatment.
  * One session of microneedling using derma roller 1.5 mm will be done.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment (Experimental): microneedling.
  Interventions: Procedure: Microneedling
- No treatment (No Intervention): No treatment will be done to these hypopigmented lesions

INTERVENTIONS:
Procedure: Microneedling — One session of microneedling will be performed by using dermaroller 1.5 mm. The microneedling done from the edge of the normal skin towards the center of the hypopigmented lesion in all the directions (horizontal, vertical. diagonal).
  Arms: treatment

SUMMARY:
Acquired hypomelanosis is a type of cutaneous melanocytopenic hypomelanosis, denoting the lightening of the skin due to a reduction in the number of epidermal and/or follicular melanocytes secondary to physical agents,post-inflammatory, and iatrogenic (steroids).

Derma roller is the basic device of microneedling , performs superficial, controlled puncturing of the skin by rolling with miniature fine needles and used as a collagen induction therapy and a transdermal delivery system for therapeutic drugs and vaccines.

This minute trauma to the skin that activates regenerative mechanisms and wound healing by releasing growth factors. The release of cytokines and deposition of hemosiderin from dermal bleeding induce the activation of melanocyte and stimulate skin pigmentation plus transdermal traveling of melanocyte

DETAILED DESCRIPTION:
The aim of this study to evaluate the efficacy and safety of microneedling as a treatment model for patients with acquired hypomelanosis.

Patients with an acquired hypomelanosis from outpatient clinic, department of dermatology, Cairo university,n=20. including:

▪Patients, both genders and older than 18 years with localized acquired hypomelanosis

Excluding:

* Congenital and hereditary hypomelanosis.
* Vitiligo
* Pregnancy and lactation.
* Patients with a history of any autoimmune disease.
* Patients with a history of keloid formation.
* Patient on systemic steroids, retinoids, immunosuppressant or anticoagulant therapy.

Methodology in details:

* An informed written consent will be obtained from the patient or his legal guardian if he is younger than 21years old.
* For every patient detailed history will focus on the onset, course, duration of hypomelanosis, the type of insult, previous treatments, systemic illness and drug history. The examination will describe the anatomical site, size, degree of skin lightening, skin texture and presence or absence of hair in the affected area.
* The area to be treated will be specified and split into two halves then randomized into one of both arms: treatment or no treatment.
* One session of microneedling will be performed on the treatment arm by using dermaroller 1.5 mm long. The microneedling will be done from the edge of the normal skin towards the center of the hypopigmented lesion in all the directions (horizontal, vertical. diagonal).
* Patients will be then monitored for three months for signs of repigmentation.
* Patient's improvement will be objectively assessed monthly for repigmentation using patient's and physician's scales.

Possible Risk:

Pain, transient bleeding, erythema, mild edema and infection at the site of microneedling. Failure of treatment is also a possibility.

Primary outcomes:

Efficacy of microneedling for acquired hypomelanosis after 3 months.

Secondary outcome:

Safety as defined by the occurrence of adverse events during, shortly after the procedure (2weeks), and after 3 months.

Sample size(number of patients included):20 patients

Source of funding: self funding

ELIGIBILITY:
Inclusion Criteria:

* Localized acquired hypomelanosis secondary to any insult, post-inflammatory or iatrogenic of no more than 2 years duration, affecting any anatomical site except genitalia, of any size larger than 3 cm in diameter.
* Patients older than 18 years old, consenting to go through the microneedling procedure.
* Both genders.

Exclusion criteria:

* Congenital and hereditary hypomelanosis.
* Vitiligo
* Pregnancy and lactation.
* Patients with history of any autoimmune disease.
* Patients with history of keloids formation.
* Patient on systemic steroids, retinoids, immunosuppressant or anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of microneedling for acquired hypomelanosis assessed by skin mapping for peripheral tanning. | 3 months post treatment
  drawing the lesion's surface area through transparent stencil paper
Efficacy of microneedling for acquired hypomelanosis assessed by visual analogue scale for surface tanning | 3 months post treatment
  using hue skin tone color scale
Efficacy of microneedling for acquired hypomelanosis assessed by vitiligo extent score for a target area for marginal and perifollicular repigmentation. | 3 months post treatment
  The repigmentation assessed by percentage value range from 0- 100% where the 100 % means full repigmentation, the value is a result of an equation where the estimated percentage of marginal repigmentation add to ( remaining area (%) plus estimated percent of perifollicular pigmentation in the remaining area(%) divided by 100)
Efficacy of microneedling for acquired hypomelanosis assessed by the patient's satisfaction score | 3 months post treatment
  3-point scale (not satisfied, moderately satisfied, extremely satisfied).
Efficacy of microneedling for acquired hypomelanosis assessed by patient global percent of his own improvement(0-100%). | 3 months post treatment
  the patient evaluation to lesion by percentage value for repigmentation ranged from 0- 100% which represent full repigmentation.
Efficacy of microneedling for acquired hypomelanosis assessed by mean physician's global assessment for percent of improvement (0-100%). | 3 moonths post treatment.
  One unblinded and 2 blinded investigators assessed the global improvement through photographs of the lesions before and after 3 months of therapy. The lesions were photographed on a black background using a single reflex camera with standardized settings (ambient light, same position, and distance from the patient).

SECONDARY OUTCOMES:
Incidence of microneedling adverse events | Day 1 to 14 and after 3 months.
  Safety as defined by occurrence of pain, bleeding, local infection, skin flaking, and scarring during, shortly after the procedure (2weeks), and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled H El-Hoshy, MD, Principal Investigator — Professor of Dermatology,Cairo University; Vanessa G Hafez, MD, Principal Investigator — Associate Professor of Dermatology, Cairo University; Julbahar M Ibrahim, M.B.,B.CH, Principal Investigator — Dermatology Resident
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeitlin RE. Long-term psychosocial sequelae of paediatric burns. Burns. 1997 Sep;23(6):467-72. doi: 10.1016/s0305-4179(97)00045-4. PMID 9429023
- [Background] Tyack ZF, Pegg S, Ziviani J. Postburn dyspigmentation: its assessment, management, and relationship to scarring--a review of the literature. J Burn Care Rehabil. 1997 Sep-Oct;18(5):435-40. doi: 10.1097/00004630-199709000-00012. PMID 9313126
- [Background] Sperry K. Tattoos and tattooing. Part I: History and methodology. Am J Forensic Med Pathol. 1991 Dec;12(4):313-9. doi: 10.1097/00000433-199112000-00008. PMID 1807141
- [Background] Singh A, Yadav S. Microneedling: Advances and widening horizons. Indian Dermatol Online J. 2016 Jul-Aug;7(4):244-54. doi: 10.4103/2229-5178.185468. PMID 27559496
- [Background] Siadat AH, Rezaei R, Asilian A, Abtahi-Naeini B, Rakhshanpour M, Raei M, Hosseini SM. Repigmentation of Hypopigmented Scars Using Combination of Fractionated Carbon Dioxide Laser with Topical Latanoprost Vs. Fractionated Carbon Dioxide Laser Alone. Indian J Dermatol. 2015 Jul-Aug;60(4):364-8. doi: 10.4103/0019-5154.160481. PMID 26288404
- [Background] Kahn AM, Cohen MJ. Treatment for depigmentation following burn injuries. Burns. 1996 Nov;22(7):552-4. doi: 10.1016/0305-4179(96)88885-1. PMID 8909758
- [Background] Imokawa G. Autocrine and paracrine regulation of melanocytes in human skin and in pigmentary disorders. Pigment Cell Res. 2004 Apr;17(2):96-110. doi: 10.1111/j.1600-0749.2003.00126.x. PMID 15016298
- [Background] Hou A, Cohen B, Haimovic A, Elbuluk N. Microneedling: A Comprehensive Review. Dermatol Surg. 2017 Mar;43(3):321-339. doi: 10.1097/DSS.0000000000000924. PMID 27755171
- [Background] Glaich AS, Rahman Z, Goldberg LH, Friedman PM. Fractional resurfacing for the treatment of hypopigmented scars: a pilot study. Dermatol Surg. 2007 Mar;33(3):289-94; discussion 293-4. doi: 10.1111/j.1524-4725.2007.33058.x. PMID 17338685
- [Background] Cho S, Zheng Z, Park YK, Roh MR. The 308-nm excimer laser: a promising device for the treatment of childhood vitiligo. Photodermatol Photoimmunol Photomed. 2011 Feb;27(1):24-9. doi: 10.1111/j.1600-0781.2010.00558.x. PMID 21198879
- [Background] Chadwick S, Heath R, Shah M. Abnormal pigmentation within cutaneous scars: A complication of wound healing. Indian J Plast Surg. 2012 May;45(2):403-11. doi: 10.4103/0970-0358.101328. PMID 23162241
- [Background] Busch KH, Bender R, Walezko N, Aziz H, Altintas MA, Aust MC. Combination of medical needling and non-cultured autologous skin cell transplantation (ReNovaCell) for repigmentation of hypopigmented burn scars. Burns. 2016 Nov;42(7):1556-1566. doi: 10.1016/j.burns.2016.04.009. Epub 2016 May 4. PMID 27156803
- [Background] Busch KH, Bender R, Walezko N, Aziz H, Altintas MA, Aust MC. Combination of medical needling and non-cultured autologous skin cell transplantation (renovacell) for repigmentation of hypopigmented burn scars in children and young people. Ann Burns Fire Disasters. 2016 Jun 30;29(2):116-122. PMID 28149233
- [Background] Aust MC, Fernandes D, Kolokythas P, Kaplan HM, Vogt PM. Percutaneous collagen induction therapy: an alternative treatment for scars, wrinkles, and skin laxity. Plast Reconstr Surg. 2008 Apr;121(4):1421-1429. doi: 10.1097/01.prs.0000304612.72899.02. PMID 18349665
- [Background] Alexiades-Armenakas MR, Bernstein LJ, Friedman PM, Geronemus RG. The safety and efficacy of the 308-nm excimer laser for pigment correction of hypopigmented scars and striae alba. Arch Dermatol. 2004 Aug;140(8):955-60. doi: 10.1001/archderm.140.8.955. PMID 15313811
- [Background] Acikel C, Ulkur E, Guler MM. Treatment of burn scar depigmentation by carbon dioxide laser-assisted dermabrasion and thin skin grafting. Plast Reconstr Surg. 2000 May;105(6):1973-8. doi: 10.1097/00006534-200005000-00009. PMID 10839394
- [Derived] Elhoshy K, Ibrahim J, Hafez V. Microneedling in Localized Acquired Hypomelanosis: A Randomized Controlled Trial. Dermatol Surg. 2025 Mar 1;51(3):257-262. doi: 10.1097/DSS.0000000000004447. Epub 2024 Nov 25. PMID 39584682